CLINICAL TRIAL: NCT00881855
Title: Comparative, Randomized, Single-Dose, 2-way Crossover Bioavailability Study of Sandoz GmbH and Bristol-Myers Squibb (Cefzil) 500 mg Cefprozil Tablets In Healthy Adults Volunteers Under Fed Conditions.
Brief Title: To Demonstrate the Relative Bioavailability of Cefzil 500 mg Cefprozil Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AA17501
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2009-04

CONDITIONS: Healthy
Keywords: Antibiotics
MeSH Terms: interventions — Cefprozil

ARMS (2):
- 1 (Experimental): Cefprozil 500 mg Tablets (Sandoz, GmbH)
  Interventions: Drug: Cefprozil 500 mg Tablets (Sandoz, GmbH)
- 2 (Active Comparator): Cefzil (Cefprozil) 500 mg Tablets (Bristol-Myers Squibb, USA)
  Interventions: Drug: Cefzil (Cefprozil) 500 mg Tablets (Bristol-Myers Squibb, USA)

INTERVENTIONS:
Drug: Cefprozil 500 mg Tablets (Sandoz, GmbH)
  Arms: 1
Drug: Cefzil (Cefprozil) 500 mg Tablets (Bristol-Myers Squibb, USA)
  Arms: 2

SUMMARY:
The purpose of this study is to Demonstrate the Relative Bioavailability of Cefzil 500 mg Cefprozil Tablets Under Fed Conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2004-03; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Morelli, M.D., Principal Investigator — MDS Pharma Services